CLINICAL TRIAL: NCT04131660
Title: Efficacy of Volume Targeted Pressure Support Ventilation vs. Pressure Support Ventilation in Patients With Acute Respiratory Failure at Risk of Obstructive Apneas or Obesity Hypoventilation
Brief Title: Efficacy of Volume Ventilation in Patients With Acute Respiratory Failure at Risk of Obstructive Apneas or Obesity Hypoventilation
Acronym: VONIVOO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/409/HP
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Acute Respiratory Failure; Hypercapnic Respiratory Failure; Respiratory Acidosis; Obesity; Hypoventilation Syndrome; Apnea, Obstructive
Keywords: non-invasive ventilation; respiratory failure; obese; obesity; Hypoventilation Syndrome; apnea; hypercapnic; acidosis; AVAPS-AE; VONIVOO
MeSH Terms: conditions — Respiratory Insufficiency; Acidosis, Respiratory; Obesity; Sleep Apnea, Obstructive; Apnea; Hypercapnia; Acidosis

STUDY DESIGN:
Intervention Model Description: The patients are randomized in 2 arms at their admission :
  * S/T mode arm : the patient is ventilated as the standard procedure of the ICU, with settings defined by the pratician.
  * AVAPS-AE mode arm : the pratician sets NIV with a positive expiratory pressure set between 4 and 14 cmH2O, an inspiratory support between 14 and 24 cmH2O and a target tidal volume between 8 and 10 mL/kg of an ideal weight (Size (m) * Size (m) * 23).
Who Masked: Participant
Masking Description: The ventilator used in both arms will be similar in appareance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AVAPS-AE mode (Experimental): A volume targeted pressure support ventilation mode
  Interventions: Device: AVAPS-AE mode during NIV
- S/T mode (Active Comparator): A pressure support ventilation mode
  Interventions: Device: S/T mode during NIV

INTERVENTIONS:
Device: AVAPS-AE mode during NIV — NIV will be setup in AVAPS-AE mode, with a Trilogy ventilation device (Respironics, Murrysville, PA). The range of positive expiratory pressure will be set between 4 and 14 cmH2O. The range of inspiratory pressure support will be set between 14 and 24 cmH2. The target tidal volume will be set to achieve 8 to 10 mL/kg of ideal body weight (Size (m) * Size (m) * 23).
  Arms: AVAPS-AE mode
Device: S/T mode during NIV — NIV will be setup in ST mode, with a Trilogy ventilation device (Respironics, Murrysville, PA).
  The physician will decide the level of positive expiratory pressure and of pressure support.
  Arms: S/T mode

SUMMARY:
This study compares a volume targeted pressure support non-invasive ventilation with an automatic PEP regulation (AVAPS-AE mode) to a pressure support non-invasive ventilation (S/T mode) in patients with acute hypercapnic respiratory failure with acidosis. This study focuses on patients at risk of obstructive apneas or obesity-hypoventilation syndrom (BMI≥30 kg/m²). Half of participants (33 patients) will receive non invasive ventilation with AVAPS-AE mode, the other half will receive non-invasive ventilation with S/T mode.

DETAILED DESCRIPTION:
So far, in respiratory intensive care units, the usual treatment of patients with acute hypercapnic respiratory failure with acidosis is non-invasive ventilation set with a pressure support mode (S/T or VS/AI mode depending on the ventilator manufacturer).

AVAPS-AE mode is a volume targeted pressure support mode with an automatic PEP. With the forced oscillations method, the ventilator is able to detect the obstruction and the resistances of upper airways.

It allows the ventilator to change its pressure settings to keep the targeted volume and avoid apneas and hypoventilation.

That is why in patients with a BMI > 30 kg/m², at risk of obesity hypoventilation syndrom or obstructive apneas, this ventilation mode may be interesting.

AVAPS-AE has been evaluated in the home ventilation showing it is as efficient as S/T mode in controlling PaCO2.

However it has never been compared to S/T mode in acute respiratory failure care.

ELIGIBILITY:
Inclusion Criteria:

* Patient of age
* Patient benefitting of social security
* Informed patient who signed the information note and the research enlighted consent form
* Admission in respiratory intensive care unit for an acid-hypercapnic exacerbation (defined by pH≤ 7,35)
* BMI ≥ 30kg/m2
* PaCO2 > 6.5 kPa on blood gases at ICU admission

Exclusion Criteria:

* Confirmed COPD with a spirometry (VEMS/CVF < 70%)
* Pregnant women, or breast-feeding women
* Patient with a judiciary or administrative liberty deprivation
* Patients under guardianship
* Contraindication to NIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Resolution of hypercapnia | through study completion, an average of 1 year
  Time between admission and resolution of hypercapnia (≤ 6.5 kPa)

SECONDARY OUTCOMES:
Comparison of persistent apneic events on NIV (/h) during the first night | through study completion, an average of 1 year
  Comparison of persistent apneic events on NIV (/h) during the first night (determined with a respiratory polygraph) between S/T mode arm and AVAPS-AE mode arm (determined with an oxymeter)
Comparison of patient-ventilator asynchronisms during NIV (/h) | through study completion, an average of 1 year
  Comparison of patient-ventilator asynchronisms during NIV (/h) between S/T mode arm and AVAPS-AE mode arm (determined with ventilator datas and a respiratory polygraph)
Comparison of time during NIV with a oxygen saturation below 90% | through study completion, an average of 1 year
  Comparison of time during NIV with a oxygen saturation below 90% between S/T mode arm and AVAPS-AE mode arm (determined with an oxymeter)
Comparison of NIV confort | through study completion, an average of 1 year
  Comparison of NIV confort between S/T mode arm and AVAPS-AE mode arm (NIV confort determined by a visual scale: 0: very comfortable to 10:not comfortable at all)
Comparison of length of stay | through study completion, an average of 1 year
  Comparison of length of stay between S/T mode arm and AVAPS-AE mode arm

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Cuvelier, MD, PhD, Study Director — UH Rouen
Locations (1):
- CHU Rouen, Rouen, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be avaible by Email request to Dr. Patout Maxime
Supporting Information: Study Protocol, ICF
Time Frame: Within 2 years of study publication
Access Criteria: Researchers in the field of acute/chronic respiratory failure.